CLINICAL TRIAL: NCT04173598
Title: Study of the Effectiveness of a Guided Compensatory Cognitive Remediation Program for Family Caregivers in Schizophrenia: a Randomized Pilot Study
Brief Title: Cognitive Remediation Program for Family Caregivers in Schizophrenia
Acronym: CIRCUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL18_0427
Record Dates: First submitted 2019-07-19; First posted 2019-11-22 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; remediation; cognitive
MeSH Terms: conditions — Schizophrenia | interventions — Caregivers

STUDY DESIGN:
Intervention Model Description: Comparative, prospective, randomized, study including two groups of (patient / caregiver) dyads:
  * An intervention group consisting of a dyad (patient + family carer) benefiting in addition to the usual treatment from the intervention for the family carer.
  * a group consisting of a dyad (patient + caregiver) with usual care (control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): An intervention group consisting of a dyad (patient + family carer) benefiting in addition to the usual treatment from the intervention for the family carer.
  Interventions: Behavioral: Cognitive Adaptation Training for Caregivers (CAT Famille)
- Control Group (Active Comparator): A group consisting of a dyad (patient + caregiver) with usual care (control group)
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Cognitive Adaptation Training for Caregivers (CAT Famille) — Family CAT manual, with a module each week to be read according to the patient's objectives and a 15-minute webcam feedback by the psychologist.
  Arms: Intervention Group
Behavioral: Usual Care — Psycho-education manual, with a weekly reading module and a 15-minute webcam feedback by the psychology student.
  Arms: Control Group

SUMMARY:
Cognitive impairments are extremely common in schizophrenia and strongly predict deficit in daily functioning, the poor managing medication and multiple hospitalizations. Cognitive remediation is recognized to have an impact on cognitive impairments by engaging preserved cognitive functions or by implementing environmental supports that sustain independent living.

Pr. Velligan (University of San Antonio) developed and tested a manualized intervention, called Cognitive Adaptation Training. In this program, trained mental health specialists implement compensatory technique such as environmental supports in the individual's living environment to live more independently and achieve greater self-sufficiency.

However, implementing this program needs a lot of professionals and time to maintain CAT effects. This type of intervention is not often done in community care and explains the large number of patients who are dependent on family members for daily living activities. Training family members in this form of intervention would be an appropriate way to resolve these issues. Families expressed a real interest in these types of home-support strategies that CAT offers. Recently, Pr. Kidd and Pr. Velligan developed a CAT version for families and created a manual accessible to people without any knowledge of cognitive deficit. This manual helps families to select specific cognitive-adaptative strategies with their relative to achieve targeted goals. Thism ethod has been translated in French.

The aim of this study was to examine whether Web-based family Cognitive Adaptation Training can improve functioning, medication adherence and negative symptoms for individuals with schizophrenia and reduce burden for family members.

A total of 60 Dyads consisting of one caregiver and one supported individual with schizophrenia will be randomized to either a Web-based family Cognitive Adaptation Training or an Internet-based control condition. Primary outcome measured will be the score on the life skills profile. Secondary outcomes will include the global score of the Zarit burden Interview, PANSS negative score, and medication adherence.

This type of intervention is expected to be developed in territorial area where professionals are not trained to cognitive remediation and therefore substantially lowers the barrier to the deployment of cognitive intervention with other psychosocial interventions for individual with schizophrenia and their caregivers.

DETAILED DESCRIPTION:
Context and justification It has been shown that when patient's family commits to a psycho-educational programme, the relapse rate of the patients themselves is halved to an equivalent level to that of drug treatment. Cognitive disorders affect 80% of patients with schizophrenia and have deleterious consequences on their autonomy and daily functioning. Cognitive remediation has now clearly demonstrated its effectiveness in the management of these cognitive disorders, particularly with regard to compensatory approaches that aim modifying the environment and providing external support. However, access to cognitive remediation remains extremely limited. It is only available in a limited number of specialized centres. In order to allow a better access to these cognitive remediation methods and to maintain its effects over time, the objective of this research project is to develop a web-based intervention, the Cognitive Adaptative Training for Caregivers ("CAT famille"), aimed at accompanying and guiding family carers via an internet video chat with a psychologist to implement cognitive remediation techniques of compensatory approach directly into their sick relative living home.

Main and secondary objectives The main objective is to evaluate the impact of a web-based intervention aimed at training a family caregiver in cognitive remediation techniques using a compensatory approach on the daily life functioning of his/her family member suffering from schizophrenia. Secondary objectives are to assess improvement in: 1) caregiver burden, 2) caregiver and patient quality of life, 3) negative symptoms, and 4) patient compliance.

Methodology This is a comparative, prospective, randomized study including two groups of (patient/caregiver) dyads: 1) an intervention group consisting of a (patient + family carer) dyad benefiting, in addition to the usual treatment, from the intervention for the family carer, and 2) a group consisting of a (patient + caregiver) dyad with usual care (control group).

Control group: Psycho-education manual, with a weekly reading module and a 15-minute webcam feedback by the psychologist.

Intervention group: Family CAT manual, with a module each week to be read according to the patient's objectives and a 15-minute webcam feedback by the psychologist.

For all groups:

Before intervention: Neuropsychological assessment + home assessment of the environment and the performance of daily living activities by psychologist A.

After intervention: Home assessment of the environment and the performance of daily living activities by psychologist B.

The inclusion criteria are: 1) for patients: patients with schizophrenia, aged 18 to 50, who can read, understand and speak French, 2) for parents: understand, speak and read French. The main outcome will be the assessment of the patient's daily life functioning as measured by the Life Skills Profile.

Process:

Total number of visits and follow-up: 3 visits during a prospective follow-up over 10 months Duration of inclusions: 18 months and duration of statistical analysis/valuation: 3-6 months

Feasibility:

The University Service of Adult Psychiatry of the University Hospital of Montpellier is one of the schizophrenia expert centres of the Fondamental network. SUPA has proven expertise in the field of cognitive remediation (see PRME Grecco in progress). SUPA works in collaboration with the family carers of people diagnosed with schizophrenia, in particular through the Profamille program (psychoeducation for carers) and UNAFAM.

Outcomes / Perspectives:

The management of cognitive disorders is essential in the care of patients with schizophrenia, in combination with other types of therapies. This research, aimed at training family carers in the use of compensatory cognitive remediation techniques that require little knowledge of neuropsychology, will be of direct benefit to patients. The expected results will contribute to the optimization of management by demonstrating that intervention and training of relatives in compensatory cognitive techniques will improve functional autonomy.

ELIGIBILITY:
Inclusion Criteria:

-

Patient group :

* Age ≥ 18 years old and < 50 years old
* patients with a diagnosis of schizophrenia according to the criteria of DSM 5 after evaluation by the investigating psychiatrist during the preliminary medical examination
* patients who can understand, speak and read French
* Patient who has given written informed consent to participate in the study, as well as written consent from the guardian for patients under guardianship, and/or from the trusted person for patients hospitalized in Third Party Request Psychiatric Care, Psychiatric Care at the request of a state representative and in a care program. If the patient is under curatorship, the curator will be informed of the study.
* Subject's participation in the study noted in the medical file
* Obligation to be a member or beneficiary of a social security scheme

Family caregiver group :

* The family carer is actively involved in the care of his or her relative with schizophrenia assessed by having at least one contact per week with the patient (Kidd et al., 2016).
* The carer has an internet connection with a video chat application
* Be under 75 years of age
* Understand, read and speak French
* Having signed an informed consent form
* Obligation to be a member or beneficiary of a social security scheme The exclusion period during which recruited patients cannot be included in another protocol is one day after the end of the evaluations. This is specified on the consent form.

Exclusion Criteria:

-

Patient group :

* Patients with a history of severe head injury and/or neurological pathology with cognitive impact.
* Patient who has benefited from individual or group cognitive remediation.

Family caregiver group :

* dementia diagnosis
* a history of neurological pathology (epilepsy, multiple sclerosis, parkinson's disease, amyotrophic lateral sclerosis, Huntington's disease)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Life Skills Profile Score (LSP-39) | Baseline
  The "Life Scale Profile" (LSP), validated in French by Mohr et al (2004), is a scale used to assess the subject's life skills profile, particularly for patients with schizophrenia. It is a hetero-questionnaire based on the patient's functioning during the last week (excluding the acute or relapse phase). The scale is composed of 20 items picked-up in an ensemble of 39 questions. The instruction is to rate each item on a scale from 1 to 4: "always, usually, rarely and never". The lower the score, the more the patient has a deficit profile in terms of life. The maximum score is 80. The LSP scale assesses 5 subscores of life skills: sociability, self-management, treatment compliance, antisocial behaviours and strange behaviours. The total duration of the test is about 30 minutes.
Life Skills Profile Score (LSP-39) | 16 weeks
  The "Life Scale Profile" (LSP), validated in French by Mohr et al (2004), is a scale used to assess the subject's life skills profile, particularly for patients with schizophrenia. It is a hetero-questionnaire based on the patient's functioning during the last week (excluding the acute or relapse phase). The scale is composed of 20 items picked-up in an ensemble of 39 questions. The instruction is to rate each item on a scale from 1 to 4: "always, usually, rarely and never". The lower the score, the more the patient has a deficit profile in terms of life. The maximum score is 80. The LSP scale assesses 5 subscores of life skills: sociability, self-management, treatment compliance, antisocial behaviours and strange behaviours. The total duration of the test is about 30 minutes.
Life Skills Profile Score (LSP-39) | 6 months
  The "Life Scale Profile" (LSP), validated in French by Mohr et al (2004), is a scale used to assess the subject's life skills profile, particularly for patients with schizophrenia. It is a hetero-questionnaire based on the patient's functioning during the last week (excluding the acute or relapse phase). The scale is composed of 20 items picked-up in an ensemble of 39 questions. The instruction is to rate each item on a scale from 1 to 4: "always, usually, rarely and never". The lower the score, the more the patient has a deficit profile in terms of life. The maximum score is 80. The LSP scale assesses 5 subscores of life skills: sociability, self-management, treatment compliance, antisocial behaviours and strange behaviours. The total duration of the test is about 30 minutes.

SECONDARY OUTCOMES:
Global score of the Zarit burden interview | Baseline
  Zarit's burden scale (Zarit et al., 1980; Hébert et al., 1993 for the French version) is a 22-item self-questionnaire measuring the burden experienced by a caregiver of an individual with a chronic disorder. The total score, which is the sum of the scores obtained for each of 22 items, varies from 0 to 88; a score less than or equal to 20 indicates a low or zero load; a score between 21 and 40 indicates a low load; a score between 41 and 60 indicates a moderate load; a score greater than 60 indicates a high load.
Global score of the Zarit burden interview | 16 weeks
  Zarit's burden scale (Zarit et al., 1980; Hébert et al., 1993 for the French version) is a 22-item self-questionnaire measuring the burden experienced by a caregiver of an individual with a chronic disorder. The total score, which is the sum of the scores obtained for each of 22 items, varies from 0 to 88; a score less than or equal to 20 indicates a low or zero load; a score between 21 and 40 indicates a low load; a score between 41 and 60 indicates a moderate load; a score greater than 60 indicates a high load.
Global score of the Zarit burden interview | 6 months
  Zarit's burden scale (Zarit et al., 1980; Hébert et al., 1993 for the French version) is a 22-item self-questionnaire measuring the burden experienced by a caregiver of an individual with a chronic disorder. The total score, which is the sum of the scores obtained for each of 22 items, varies from 0 to 88; a score less than or equal to 20 indicates a low or zero load; a score between 21 and 40 indicates a low load; a score between 41 and 60 indicates a moderate load; a score greater than 60 indicates a high load.
Patient quality of life: S-QoL 18 | Baseline
  The quality of life of patients is assessed by the Quality of Life Scale (S-QoL 18) is a shortened version of the S-QoL 41 scale whose validity and psychometric properties have been validated in patients with schizophrenia. The self-administered questionnaire assesses the impact of patients' difficulties on their quality of life through 8 dimensions: psychological well-being, self-esteem, family relationships, friendly relationships, resilience, physical well-being, autonomy and emotional life. The duration of the test is 7 minutes.
Patient quality of life: S-QoL 18 | 16 weeks
  The quality of life of patients is assessed by the Quality of Life Scale (S-QoL 18) is a shortened version of the S-QoL 41 scale whose validity and psychometric properties have been validated in patients with schizophrenia. The self-administered questionnaire assesses the impact of patients' difficulties on their quality of life through 8 dimensions: psychological well-being, self-esteem, family relationships, friendly relationships, resilience, physical well-being, autonomy and emotional life. The duration of the test is 7 minutes.
Patient quality of life: S-QoL 18 | 6 months
  The quality of life of patients is assessed by the Quality of Life Scale (S-QoL 18) is a shortened version of the S-QoL 41 scale whose validity and psychometric properties have been validated in patients with schizophrenia. The self-administered questionnaire assesses the impact of patients' difficulties on their quality of life through 8 dimensions: psychological well-being, self-esteem, family relationships, friendly relationships, resilience, physical well-being, autonomy and emotional life. The duration of the test is 7 minutes.
Caregiver quality of life: S-QoL 18 | Baseline
  The quality of life of caregivers is assessed by the Quality of Life Scale: As for patients, we will use the Quality of Life Scale (S-QoL 18). The self-administered questionnaire assesses the impact of patients' difficulties on their quality of life through 8 dimensions: psychological well-being, self-esteem, family relationships, friendly relationships, resilience, physical well-being, autonomy and emotional life. The duration of the test is 7 minutes.
Caregiver quality of life: S-QoL 18 | 16 weeks
  The quality of life of caregivers is assessed by the Quality of Life Scale: As for patients, we will use the Quality of Life Scale (S-QoL 18). The self-administered questionnaire assesses the impact of patients' difficulties on their quality of life through 8 dimensions: psychological well-being, self-esteem, family relationships, friendly relationships, resilience, physical well-being, autonomy and emotional life. The duration of the test is 7 minutes.
Caregiver quality of life: S-QoL 18 | 6 months
  The quality of life of caregivers is assessed by the Quality of Life Scale: As for patients, we will use the Quality of Life Scale (S-QoL 18). The self-administered questionnaire assesses the impact of patients' difficulties on their quality of life through 8 dimensions: psychological well-being, self-esteem, family relationships, friendly relationships, resilience, physical well-being, autonomy and emotional life. The duration of the test is 7 minutes.
Negative symptoms | Baseline
  Clinical Assessment Interview for Negative symptoms (CAINS) (Kring et al., 2013). CAINS is a recently developed tool to evaluate the 2 dimensions of negative symptomatology highlighted in the literature, i.e. the motivation dimension and the decreased emotional expressivity dimension. It has been translated into French by our team (Raffard et al., currently under validation). It includes 13 items (9 for the amotivation dimension and 4 for the expressivity dimension) evaluated during a semi-structured interview.
Negative symptoms | 6 months
  Clinical Assessment Interview for Negative symptoms (CAINS) (Kring et al., 2013). CAINS is a recently developed tool to evaluate the 2 dimensions of negative symptomatology highlighted in the literature, i.e. the motivation dimension and the decreased emotional expressivity dimension. It has been translated into French by our team (Raffard et al., currently under validation). It includes 13 items (9 for the amotivation dimension and 4 for the expressivity dimension) evaluated during a semi-structured interview.
Patient compliance | Baseline
  Medication Adherence Rating Scale (Misdrahi et al., 2004). This scale is one of the most widely used tools to assess compliance in individuals with schizophrenia. This is a self-administered questionnaire with 10 yes/no items offering a total score from 0 (low compliance) to 10 (high compliance).
Patient compliance | 16 weeks
  Medication Adherence Rating Scale (Misdrahi et al., 2004). This scale is one of the most widely used tools to assess compliance in individuals with schizophrenia. This is a self-administered questionnaire with 10 yes/no items offering a total score from 0 (low compliance) to 10 (high compliance).
Patient compliance | 6 months
  Medication Adherence Rating Scale (Misdrahi et al., 2004). This scale is one of the most widely used tools to assess compliance in individuals with schizophrenia. This is a self-administered questionnaire with 10 yes/no items offering a total score from 0 (low compliance) to 10 (high compliance).

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Raffard, PU, Principal Investigator — CHU Montpellier (s-raffard@chu-montpellier.fr)
Locations (1):
- Service Universitaire de psychiatrie adulte, Montpellier, France